CLINICAL TRIAL: NCT04438668
Title: Evaluation of the Safety and Performance of Centaflow as a Routine Assessment of Placental Vascular Function and Foetal Cardiovascular Health
Brief Title: Evaluation of the Safety and Performance of Centaflow
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centaflow (Industry)
Collaborators: Rigshospitalet, Denmark (Other); Viborg Regional Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 2019-01
Record Dates: First submitted 2020-06-08; First posted 2020-06-19 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2021-12

CONDITIONS: Fetal Growth Restriction
MeSH Terms: conditions — Fetal Growth Retardation

STUDY DESIGN:
Intervention Model Description: Randomised Controlled Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (Active Comparator): Standard care (SC) for screening for FGR is a healthcare provider auscultating the foetal heart rate with a standard stethoscope, palpation of foetal size by hand, and measuring the size of the woman's uterus with a tape measure, and comparing the measurement to the expected measurement for the gestational age of the foetus.
  Interventions: Diagnostic Test: Standard Care
- Standard Care and Centaflow (Experimental): Centaflow uses sound-derived maternal intra-arterial turbulence as a marker of foetal growth restriction (FGR) and provides information on the foetal heart rate. Indication for use is as a screening device for FGR in women beyond 27 weeks of pregnancy with a singleton pregnancy.
  Interventions: Device: Centaflow and Standard Care

INTERVENTIONS:
Device: Centaflow and Standard Care — The intervention is screening methods
  Other Names: Standard Care is Symphysis-fundal measure and fetal weight estimation
  Arms: Standard Care and Centaflow
Diagnostic Test: Standard Care — The intervention is screening methods
  Other Names: Symphysis-fundal measure and fetal weight estimation
  Arms: Standard Care

SUMMARY:
The aim of this study is to evaluate the safety and performance of an acoustic approach based on skin-contact microphones as a routine assessment of placental vascular function as predictor of fetal growth restriction.

DETAILED DESCRIPTION:
Evaluation of the safety and performance of Centaflow as routine antenatal assessment of placental vascular function as predictor of fetal growth restriction is performed by randomizing singleton pregnant women with ultrasound-based gestations for either standard care (SC) or SC and Centaflow (CF).

The subjects will be randomized in ratio 1:1 in both groups and examined in pregnancy weeks 27-29, 34-36 and 37-39.

ELIGIBILITY:
Inclusion Criteria

* Female subjects over the age of 18 years.
* Subejct is pregnant, carries only one fetus and has been pregnancy dated by ultrasound scan (Hadlock reference).

Exclusion Criteria

* Fetal abnormality known to affect growth, diagnosed in-utero or through 12 days postnatally.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1704 (Estimated)
Dates: Start 2020-06-03 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Fetal Growth Restriction (FGR) | At birth
  Outcome is the classification of each neonate as FGR or as non-FGR at birth. FGR is defined as birth weight below the 3rd percentile or birth weight below the 10th percentile and an antenatally detected abnormal umbilical artery blood flow.
Safety: occurrence of device-related adverse events | At gestational week 27-29
  Outcome is the occurrence of device-related adverse events and their classification as serious or not.
Safety: occurrence of device-related adverse events | At gestational week 34-36
  Outcome is the occurrence of device-related adverse events and their classification as serious or not.
Safety: occurrence of device-related adverse events | At gestational week 37-39
  Outcome is the occurrence of device-related adverse events and their classification as serious or not.

SECONDARY OUTCOMES:
Mode of delivery | At birth
  Outcome is the mode of delivery being either A) uncomplicated vaginal, B) complicated vaginal, C) planned cesarean section or D) emergency cesarean section.
Neonatal Intensive Care Unit | At 12 days postpartum
  Outcome is the occurrence of admission to the Neonatal Intensive Care Unit

CONTACTS AND LOCATIONS:
Overall Officials: Richard Farlie, MD, MI, MHM, Principal Investigator — Viborg Regional Hospital
Locations (2):
- Denmark (2):
  - Juliane Marie Centeret, Rigshospitalet, Copenhagen
  - Obstetrical Department, Regional Hospital Viborg, Viborg

IPD SHARING:
Plan to Share IPD: No
Sharing raw data is inconsistent with the ethics application form and the participant informed consent materials.